CLINICAL TRIAL: NCT02374203
Title: Clinical Dietitian, Dietetic Service, Mackay Memorial Hospital
Brief Title: Nutritional Needs and Intake on Clinical Outcomes in Mechanically Ventilated Critically Ill Elderly Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mackay Memorial Hospital (Other)
Responsible Party: Principal Investigator, Pi-Hui Hsu, Dietitian, Dietetic service, Mackay Memorial Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 14MMHIS229
Record Dates: First submitted 2014-12-11; First posted 2015-02-27 (Estimated); Last update posted 2018-09-05 (Actual); Status verified 2018-08

CONDITIONS: Critical Illness; Mechanical Ventilation; Elderly
Keywords: Indirect Calorimetry; Harris-Benedict equation; critical elderly; mNUTRIC score; high nutritional risk
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Intervention Model Description: Patients were randomized 1:1 to two tube feeding regimens: general formula and high protein formula (1.5~2.0 gm/kg BW).
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- high protein enteral nutrition (Experimental): supply protein over 1.5 gm/kg body weight
  Interventions: Dietary Supplement: high protein enteral nutrition

INTERVENTIONS:
Dietary Supplement: high protein enteral nutrition — supply protein over 1.5 gm/kg body weight

SUMMARY:
The purposes of this study were to investigate the caloric requirement and clinical outcomes in mechanically ventilated critically ill elderly patients and identify those at high nutritional risk who require high protein formula intervention.

DETAILED DESCRIPTION:
The elderly population is rapidly increasing, but studies on calorie requirement in critically ill elderly patients are few, and indirect calorimetry (IC) is not available in every intensive care unit (ICU). The aim of this study was to compare IC and Harris-Benedict (HB) predictive equation in different BMI (body mass index) groups. And to investigate whether the nutrition intake from EN (enteral nutrition) and PN (parenteral nutrition) created a better clinical outcome than EN alone in HNR (high nutritional risk) mechanically ventilated critically ill elderly patients.Inclusion criteria were: age ≧65 years old, APACHE Π score ≧15, mechanical ventilation ≧48 hours and on NG tube feeding. Nutritional risk was screened by mNUTRIC and GNRI. Indirect calorimetry and HB equation were used to assess energy requirements. Patients were randomized 1:1 to two tube feeding regimens: general formula and high protein formula (1.5~2.0 gm/kg BW). Nutritional intake from EN, the type and amount of intravenous nutrition within 7 days, tolerance to feeding, MVD (Mechanical Ventilation Day), newly diagnosed VAP (Ventilator Associated Pneumonia), ICU and hospital LOS (Length of Stay) and date of death were recorded. We used SAS version 9.4 for statistical analysis. Statistically significance was set at α=0.05.

ELIGIBILITY:
Inclusion Criteria:

* APACHE Π score ≧ 15
* ≧ 65 years
* on mechanical ventilation ≧48 hours
* received EN

Exclusion Criteria:

* Use of total parenteral nutrition
* Fasting >5 days
* Brain death
* Terminal cancer

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 190 (Actual)
Dates: Start 2014-12-26 (Actual); Primary Completion 2016-06-30 (Actual); Study Completion 2016-06-30 (Actual)

PRIMARY OUTCOMES:
Determination of the energy requirements in critically ill elderly patients | first 5 days in the ICU
  A total of 177 critically ill elderly patients (≧ 65 years old) underwent IC for measured resting energy expenditure (MREE). Estimated calorie requirement was calculated by the HB equation, using actual body weight (ABW) and ideal body weight (IBW) separately. Patients were divided into four BMI groups. One-way ANOVA and Pearson's correlation coefficient were used for statistical analyses.

SECONDARY OUTCOMES:
Higher Enteral Nutrition Intake May Reduce Hospital Mortality | first 28 days in the ICU
  We included patients ≧ 65 years on mechanical ventilation ≧ 48 hours and received EN. Nutritional status was evaluated by mNUTRIC score. We calculated the energy and protein requirements as Harris-Benedict equation ╳ 1.0~1.3 and 1.0~2.0 gm/kg body weight respectively. Nutrition intake from EN and PN was recorded within 7 days. ICU and hospital mortalities in HNR elderly patients who could achieve more or less 80% of the prescribed nutrition were compared.

CONTACTS AND LOCATIONS:
Overall Officials: Pi-Hui Hsu, Principal Investigator — Mackay Memorial Hospital
Locations (1):
- Mackay Memorial Hospital, Taipei, Taiwan

REFERENCES:
- [Background] Hsu PH, Lee CH, Kuo LK, Kung YC, Chen WJ, Tzeng MS. Higher Energy and Protein Intake from Enteral Nutrition May Reduce Hospital Mortality in Mechanically Ventilated Critically Ill Elderly Patients. International Journal of Gerontology. Available online 26 March 2018. https://doi.org/10.1016/j.ijge.2018.03.001
- [Result] Hsu PH, Lee CH, Kuo LK, Kung YC, Chen WJ, Tzeng MS. Determination of the energy requirements in mechanically ventilated critically ill elderly patients in different BMI groups using the Harris-Benedict equation. J Formos Med Assoc. 2018 Apr;117(4):301-307. doi: 10.1016/j.jfma.2017.12.010. Epub 2018 Jan 12. PMID 29336938